CLINICAL TRIAL: NCT03983837
Title: Elemental Diet for Treatment of Inflammatory Bowel Disease in Patients With Chronic Granulomatous Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190108; 19-I-0108
Record Dates: First submitted 2019-06-07; First posted 2019-06-12 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12-09

CONDITIONS: Chronic Granulomatous Disease; Inflammatory Bowel Disease
Keywords: Inflammatory Bowel Disease; Crohn disease; Ulcerative Colitis; Glucocorticoids; Microbiome
MeSH Terms: conditions — Granulomatous Disease, Chronic; Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Participants will be on this diet for 4 weeks. The amount per serving will be determined on the basis of the participant s weight and caloric needs, as determined by a staff dietician.
  Interventions: Other: Neocate Splash

INTERVENTIONS:
Other: Neocate Splash — Neocate Splash is a hypoallergenic, amino acid based elemental liquid diet that is taken orally.

SUMMARY:
Background:

Bacteria that live inside the stomach and intestines are important for health. Chronic granulomatous disease (CGD) and inflammatory bowel disease (IBD) can make people have unhealthy bacteria. This can lead to gastrointestinal (GI) problems. Researchers want to see if people with CGD and IBD feel better when they change the bacteria in the stomach by following a special liquid diet.

Objective:

To see if an elemental diet can change the bacteria in the stomach and intestines of people with CGD and IBD. Also, to see if this helps GI symptoms.

Eligibility:

People ages 8-65 years with CGD, CGD-associated colitis, and IBD.

Design:

Participants will first be screened with:

Upper GI endoscopy and/or colonoscopy. A long, thin tube with a tiny camera at the end will be passed into the participant s body through the mouth or anus. Tissue will be collected. Participants will be sedated for the procedure. They will be sedated using a special mask or small plastic tube placed in an arm vein using a needle.

Participants will be put on the special diet for up to 4 weeks. They will stay in the hospital for up to 2 weeks. They will have check-ups. They will have blood, urine, and stool samples collected. They will keep a symptom diary to record how they feel and any GI symptoms.

Participants will have 2 follow-up visits. The first will be right after they finish the diet. The second will be 4 weeks later. They will have blood, urine, and stool samples collected. They will learn about re-introducing other foods into their diet.

DETAILED DESCRIPTION:
Chronic granulomatous disease (CGD) is a rare genetic immune disorder that results in recurrent and severe infections, and inflammatory dysregulation. For almost 50% of patients with CGD, this inflammation causes severe inflammatory bowel disease (IBD). However, treatment is long term and challenging as CGD-IBD is prone to relapse, and use of immune modulators must be balanced with increased risk of infectious complications. Conventional IBD (Crohn disease and ulcerative colitis) is likely caused by an inappropriate inflammatory response to intestinal microbes, which is influenced by the environment in a genetically susceptible host. While it is not yet clear if intestinal dysbiosis is a result or cause of intestinal inflammation, studies suggest that correcting intestinal dysbiosis may improve intestinal inflammation. Studies in patients with conventional IBD suggest that strict dietary restrictions can resolve symptoms of IBD and induce remission as effectively as glucocorticoids but without the side effects of those drugs. Because these diets alter the gut microbiome, they may serve as effective treatment for CGD-IBD.

In this study, we propose to treat 5 patients >= 8 years old who have CGD and IBD with 4 weeks of an elemental diet. Participants will stay as inpatients for up to 2 weeks and will return for follow-up at the end of the diet to begin tapering off and be reintroduced to normal food. The primary objective of this study is the evaluation of changes in the microbiome before and after the elemental diet. Secondary objectives are evaluations of tolerability and safety of the diet, along with changes in local and systemic markers of inflammation, and improvement of IBD symptoms as determined by reduction in Harvey-Bradshaw Index score.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals must meet all of the following criteria to be eligible for study participation:

* Aged 8-65 years.
* Have confirmed diagnoses of CGD, CGD-associated colitis, and IBD.
* Have a Simple Endoscopic Score for Crohn Disease (SES-CD) > 3 and/or HBI >= 5.
* Able to provide informed consent.
* Willing to allow storage of biological samples for future research.
* Willing to allow genetic testing on biological samples.
* Willing to be admitted as inpatient for up to 2 weeks to initiate the elemental diet.

EXCLUSION CRITERIA:

* Pregnancy.
* Active or ongoing infection that requires antibiotics other than the participant s known prophylaxis medications.
* Any condition that, in the opinion of the investigator, contraindicates participation in this study will be excluded from study participation.

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
Change in the relative abundance of proteobacteria in stool samples obtained after elemental diet. | Day 56
  Change in the relative abundance of proteobacteria in stool samples obtained after elemental diet.

SECONDARY OUTCOMES:
Unexpected AEs possibly, probably, or definitely related to the elemental diet. | Day 0 to 56
Ability to tolerate 4 weeks of elemental diet as measured by > 75% of caloric intake via elemental diet over the 4-week period. | Day 0 to 27
Weight loss. | Day 0 to 56
Initiation of antibiotics. | Day 0 to 56
Changes in fecal calprotectin, ESR, and CRP. | Day 56
Changes in the HBI at completion of the elemental diet and at 4 weeks after completion. | Day 28 and 56
Change in alpha and beta diversity after diet | Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Christa S Zerbe, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Human data generated in this study will be shared for future research as follows:@@@-De-identified data in an NIH-funded or approved public repository.@@@-De-identified data in another public repository. @@@-Identified data in the Biomedical Translational Research Information System (automatic for activities in the CC).@@@-De-identified or identified data with approved outside collaborators under appropriate agreements.
Supporting Information: CSR
Time Frame: Data will be shared at the time of or shortly after publication.
Access Criteria: Requests for data will be reviewed and approved/disapproved by the PI.

REFERENCES:
- [Background] Jones LB, McGrogan P, Flood TJ, Gennery AR, Morton L, Thrasher A, Goldblatt D, Parker L, Cant AJ. Special article: chronic granulomatous disease in the United Kingdom and Ireland: a comprehensive national patient-based registry. Clin Exp Immunol. 2008 May;152(2):211-8. doi: 10.1111/j.1365-2249.2008.03644.x. PMID 18410635
- [Background] Magnani A, Brosselin P, Beaute J, de Vergnes N, Mouy R, Debre M, Suarez F, Hermine O, Lortholary O, Blanche S, Fischer A, Mahlaoui N. Inflammatory manifestations in a single-center cohort of patients with chronic granulomatous disease. J Allergy Clin Immunol. 2014 Sep;134(3):655-662.e8. doi: 10.1016/j.jaci.2014.04.014. Epub 2014 Jun 27. PMID 24985400
- [Background] van den Berg JM, van Koppen E, Ahlin A, Belohradsky BH, Bernatowska E, Corbeel L, Espanol T, Fischer A, Kurenko-Deptuch M, Mouy R, Petropoulou T, Roesler J, Seger R, Stasia MJ, Valerius NH, Weening RS, Wolach B, Roos D, Kuijpers TW. Chronic granulomatous disease: the European experience. PLoS One. 2009;4(4):e5234. doi: 10.1371/journal.pone.0005234. Epub 2009 Apr 21. PMID 19381301
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-I-0108.html